CLINICAL TRIAL: NCT01914640
Title: The Cross Sectional Study to Investigate the Waist Circumference Cut Off Points for the Prediction of Overweight and Obesity of the Turkish Adult Population
Brief Title: The Sex Specific Waist Circumference Cut Off Points to Predict Overweight or Obesity
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Fahri Bayram, Professor in Medicine, Faculty of the Department of Endocrinology and Metbolism, TC Erciyes University
Other Study IDs: TEMD/OBDLHT- 0001
Record Dates: First submitted 2013-07-25; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: The Focus of Study is to Determine the Waist Circumference Values to Predict Overweight or Obesity
Keywords: Waist circumference, Metabolic Syndrome, Cardiovascular risk
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adults living in Turkey: The group was enrolled from the 24 provinces of the 7 regions of Turkey. At least 3 provinces were selected from each region by a random sampling method. The populations of these 7 regions were obtained from the records of the 2000 census. The study sample included males and non-pregnant females aged between 20 and 83 years. The populations of city centers, districts, and villages were classified by using the stratified sampling method and then were selected from the data collected from the household identification forms by random sampling. The geography of Turkey was classified into three groups according to altitude. Sea level was accepted as zero. 0-300 m was taken as coastal, 300-900 m as moderate

SUMMARY:
The waist circumference (WC) cut off levels of the Caucasian people may not represent the characteristics of different ethnic groups. The investigators aimed to determine sex specific WC cut off points to predict obesity, metabolic syndrome and increased cardiovascular risk in Turkish adults.

DETAILED DESCRIPTION:
Waist circumference (WC) is an easy and reliable measure of visceral adipose tissue and a simple index of cardiovascular risk. The World Health Organization (WHO) reported sex specific WC cut off values for the Caucasian people, named as action levels 1 and 2, to define the overweight or obese people. These cut off values, originally established in a Dutch population, were later adopted by several medical organizations in order to define Metabolic Syndrome. However, these cut off levels may not necessarily represent the characteristics of the other populations. Therefore it is recommended that the sex specific WC cut off points should be established for different ethnic groups.

The investigators aimed to investigate whether the suggested sex specific WC cut off points for the Caucasian adults are appropriate for the Turkish adult population. The secondary aim of the study is to search for better WC cut off points to predict obesity, metabolic syndrome and increased cardiovascular risk in Turkish adult men and women.

ELIGIBILITY:
Inclusion Criteria:

* Adult Male or nonpregnant Female

Exclusion Criteria:

Pregnant females, Subjects younger than 20 or older than 83

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This cross-sectional study was conducted in 24 provinces from the 7 regions of Turkey. Turkish adult males and non-pregnant females were randomly enrolled from both the provincial district centers and villages, considering the demographics, economic, social, and geographical statuses.
Sampling Method: Probability Sample
Enrollment: 4310 (Actual)
Dates: Start 2003-03; Primary Completion 2004-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Waist circumference cut off levels | About a year to collect all the demographic data
  These cut off levels were determined by the receiver operating curve analyses. The sum of the highest sensitivity and specificity values of the WC levels to determine the overweight (Body mass index (BMI) > 25kg/m2) and obese (BMI>30kg/m2) adults were taken as the cut off points. The cut off points to determine the overweight, were also taken as the WC limits for the diagnosis of metabolic syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Bayram, MD. Prof., Study Director — Head of the Study Group of Hypertension, Lipid disorders and Obesity of Turkish Society of Endocrinology and Metabolism

REFERENCES:
- [Background] Gundogan K, Bayram F, Gedik V, Kaya A, Karaman A, Demir O, Sabuncu T, Kocer D, Coskun R. Metabolic syndrome prevalence according to ATP III and IDF criteria and related factors in Turkish adults. Arch Med Sci. 2013 Apr 20;9(2):243-53. doi: 10.5114/aoms.2013.34560. Epub 2013 Apr 12. PMID 23671434